CLINICAL TRIAL: NCT04889378
Title: Change of Body Composition and Functional Status Following Short-term Pre-habilitation Among Morbidly Obese Patients Before Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: National Cancer Institute, Malaysia (Other Government)
Responsible Party: Principal Investigator, HO CHIOU YI, principal investigator, Universiti Putra Malaysia
Other Study IDs: NMRR-21-355-58673
Record Dates: First submitted 2021-04-26; First posted 2021-05-17 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Short Term Pre-habilitation Before Bariatric Surgery
Keywords: obesity
MeSH Terms: conditions — Obesity | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-habilitation: participants will join prehabilitation with very low calories diet (800-1000kcal/day) and moderate intensive aerobic exercise (1 hour per section; 3 sections per day) for 2 weeks before bariatric surgery.
  Interventions: Other: prehabilitation

INTERVENTIONS:
Other: prehabilitation — very low calories diet (800-1000kcal/day) with moderate intensive aerobic exercise (1 hour per section; 3 sections per day)

SUMMARY:
Observational study is conducted in patient under short term pre-habilitation before bariatric surgery.

DETAILED DESCRIPTION:
Observational study is conducted in patient under short term pre-habilitation before bariatric surgery. Data on anthropometry (waist circumference), body compositions (weight, muscle mass, fat free mass, fat mass, fat percentage and basal metabolic rate (BMR)), and functional status (handgrips strength) are collected.

ELIGIBILITY:
Inclusion Criteria:

* Obese or severe obese patients
* Candidates for short term pre-habilitation among morbid obese patients before bariatric surgery
* Aged more than 18 years old
* Malaysian
* Provided and signed informed consent

Exclusion Criteria:

* Not a candidate for short term pre-habilitation among morbid obese patients before bariatric surgery
* Aged <18 years old
* Non-Malaysian
* Not able to provide informed consent
* chronic renal failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: morbidly obese patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
anthropometry (waist circumference in cm) | baseline and after 2 weeks
  change in waist circumference at 2 weeks
body composition (weight in kg) | baseline and after 2 weeks
  change in weight at 2 weeks. It will be measured by using BIA TANITA
body composition (muscle mass in kg) | baseline and after 2 weeks
  change in muscle mass at 2 weeks. It will be measured by using BIA TANITA
body composition (fat free mass in kg) | baseline and after 2 weeks
  change in fat free mass at 2 weeks. It will be measured by using BIA TANITA
body composition (fat mass in kg) | baseline and after 2 weeks
  change in fat mass at 2 weeks. It will be measured by using BIA TANITA
body composition (fat percentage in percentage) | baseline and after 2 weeks
  change in fat percentage at 2 weeks. It will be measured by using BIA TANITA
functional status (hand-grips strength in kg) | baseline and after 2 weeks
  change in hand-grips strength at 2 weeks. Hand-grip strength will be measured by using Jammar Dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided